CLINICAL TRIAL: NCT03186196
Title: Influence of Polymorphism C677T MTHFR and Folate Intake in Interleukins, Homocysteine and TNF-α
Brief Title: Polymorphism C677T MTHFR and Folate Intake in Inflammatory Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Jéssica Vanessa de Carvalho Lisboa, Nutritionist and Master Degree Student of Science of Nutrition, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUParaíbaaa
Record Dates: First submitted 2017-05-24; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Overweight and Obesity
Keywords: Folate; Polymorphism; Overweight and Obesity; Inflammatory markers
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Diet with 191 mcg/day of Folate
  Interventions: Dietary Supplement: Diet containing Folate
- Group 2 (Active Comparator): Diet containing 90 mcg / day of Folate
  Interventions: Dietary Supplement: Diet containing Folate

INTERVENTIONS:
Dietary Supplement: Diet containing Folate

SUMMARY:
The C677T polymorphism of the MTHFR gene is associated to several biochemicals imbalances, as changes in folic acid serum levels and some inflammatory markers, elevating the oxidative stress and increasing the risk of developing non communicable diseases (NCDs).

Thus, a diet containing folate as a main antioxidant nutrient, could reduce not only the oxidative stress, but also has many others benefits for individuals with this genetic alteration, like the anti-inflammatory function, which could help restore the altered serum levels and minimizing or avoiding the development of future diseases.

The aim of this study was to evaluate the influence of the C677T polymorphism of the MTHFR gene and the effect of a diet containing folate in the inflammatory markers levels, such as homocysteine, Tumor Necrosis Factor alpha (TNF-α) and interleukins in women with overweight or obesity. This is an intervention study, double-blind, held in a city in northeastern Brazil, with a sample of 48 adult women (20-59 years old) with BMI among 26.19 kg / m² and 49.64 kg / m². In which we evaluated the TNF-α levels, Interleukins 1β, Interleukin 6, Interleukin 8, Interleukin 12p70, Interleukin 10, homocysteine, folic acid and in addition to these markers evaluation, were made the genotyping for the C677T polymorphism in the MTHFR gene and the food consumption assessment by the 24 hour dietary recall (24HR). For the intervention, the sample was divided by randomization into two groups, each one with 24 indivuals, receiving daily during 8 weeks, a salad with 300g vegetables containing 191 ug of folate for group 1 and 90 ug for group 2.

DETAILED DESCRIPTION:
This work is linked to a population-based survey entitled "Diagnosis and Intervention II Cycle Situation Food, Nutrition and Noncommunicable Diseases prevalent over the city of João Pessoa Population / PB" (II DISANDNT / PB). For the realization of this dissertation we (teams of undergraduate researchers and graduates of Nutrition Course, masters and doctoral students of the Post Graduate Program in Nutrition Sciences (PPGCN) of UFPB) did home visits, applied questionnaires related to anthropometric and food intake assessment, by duly previously trained at the beginning of data collection and after completion of the pilot study.

After the selection of individuals from the sample of adults who participated in the II DISANDNT / JP and considering the inclusion criteria and genotyping of the C677T polymorphism in the MTHFR gene, they were invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adult women, aged 20 to 59 years old, with overweight or obesity
* Individuals of different socioeconomic conditions
* Users or not drugs
* Cognitive state preserved and accept participate

Exclusion Criteria:

* Drinkers, smokers or with neuropsychiatric disorders
* Users drugs known to interfere with the metabolism of folic acid (the last 3 months), as prednisone, hydrocortisone, dexamethasone, chloramphenicol, acetylsalicylic acid
* Multivitamin supplement users, minerals, appetite suppressants and steroids
* Individuals with chronic diseases with influence on the endocrine and metabolic system
* Pregnant or planning to become pregnant during the study period

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in value of Interleukins | 8 weeks
Change in value of homocysteine | 8 weeks

SECONDARY OUTCOMES:
Change in value of TNF-α | 8 weeks

OTHER OUTCOMES:
Change in value of folic acid | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria José de Carvalho Costa, PhD, Study Director — UFPB

IPD SHARING:
Plan to Share IPD: Yes
The data of the participants are in the excel database